CLINICAL TRIAL: NCT01561209
Title: Prospective Randomized & Controlled Study of the Role of Low Doses Amitriptyline in the Management of Chronic Neck Pain
Brief Title: Low Doses Amitriptyline & Chronic Neck Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, Dr Joseph Maarrawi, Assistant Professor : Researcher - Pain Specialist - Neurosurgeon, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMIT-CNP
Record Dates: First submitted 2012-03-14; First posted 2012-03-22 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Neck Pain
Keywords: amitryptiline; Chronic pain; Neck pain
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amitryptiline (Active Comparator): Amitryptiline 5 mg before bedtime
  Interventions: Drug: Amitryptiline
- Placebo (Placebo Comparator): Placebo pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amitryptiline — Amitryptiline 5 mg before bedtime for 2 months
  Other Names: Tryptizol; Laroxyl
  Arms: Amitryptiline
Drug: Placebo — Placebo pill
  1 before bedtime
  Other Names: No brand name
  Arms: Placebo

SUMMARY:
The objective of this prospective randomized and controlled study is to evaluate the efficacy and safety of low dose of amitriptyline (5 mg) in the management of chronic neck pain.

DETAILED DESCRIPTION:
Patients with chronic neck pain, lasting since at least 3 months, are recruited from our pain clinic. After verification of inclusion and exclusion criteria, patients consenting to enter the study are assigned randomly to one of the following groups: 1-Amitriptyline 5 mg for 2 months 2- placebo for 2 months. Co-morbidities and other painful conditions are noted, and then clinical evaluation of the patient is performed; pain is assessed according to Visual Analog Scale, anxiety, depression, insomnia and disability are evaluated by adapted scores (Bergen insomnia scale, neck pain disability score, neck pain diary & anxiety and depression score). Patients are followed at 2 months and outcome measures are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck pain (since more than 3 months, and more than 15 days/month)
* Normal neurologic exam
* X-ray = normal or loss of lordosis

Exclusion Criteria:

* Neurologic signs or symptoms
* Past history of neck surgery
* MRI = abnormal findings except for loss of lordosis
* Past cervical trauma
* severe depression
* drug abuse
* pregnancy
* Follow-up not possible
* cardiac rhythms problems
* Glaucoma
* Urinary tract obstruction or prostatism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in Visual analog scale (VAS) | 0 and 2 months after treatment
  Pain assessment on VAS at 2 months compared to baseline

SECONDARY OUTCOMES:
Change in Bergen insomnia score | 0, 2 months
  it assesses the sleep quality of the patient at 2 months compared to baseline
Change in Neck pain disability score | 0, 2 months
  NECK PAIN DISABILITY INDEX QUESTIONNAIRE at 2 months compared to baseline
side effects | Up to 12 weeks after treatment
  reporting the side effects by the patient
Percentage of satisfaction | 2 months after treatment
  Pain subjective percentage of improvement
Change in Hospital Anxiety and Depression Scale (HADS) | 0 and 2 months after treatment
  Assessment of anxiety and depressive symptoms at 2 months compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Maarrawi, MD, PhD, Principal Investigator — St Joseph University, Beirut, Lebanon
Locations (1):
- Hotel Dieu de france Hospital, Beirut, Lebanon